CLINICAL TRIAL: NCT01248728
Title: A Randomized, Placebo-Controlled Trial of Omega-3 Fatty Acids in the Treatment of Young Children With Autism
Brief Title: Omega-3 Fatty Acids For Treatment Of Young Children With Autism (OMG)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-018
Record Dates: First submitted 2010-11-22; First posted 2010-11-25 (Estimated); Results first posted 2016-05-18 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Clinical Trial; Omega-3 Fatty Acids; Toddlers
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3 Fatty Acids (Active Comparator): Children will be administered 3.75ml of the liquid formulation of Nutra Sea high-EPA (HP) (containing 1.5 gr of EPA+DHA). The starting dose will be 1.875ml (0.75 gr of EPA+DHA) and the dose will be doubled on week 2.
  Interventions: Dietary Supplement: Omega-3 Fatty Acids
- Placebo (Placebo Comparator): Children will be administered 3.75ml of the liquid formulation of Placebo. The starting dose will be 1.875ml and the dose will be doubled on week 2.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 Fatty Acids — Children will be administered 3.75ml of the liquid formulation of Nutra Sea HP (containing 1.5 gr of EPA+DHA). The starting dose will be 1.875ml (0.75 gr of EPA+DHA) and the dose will be doubled on week 2. The parents may choose to give this as a single dose or split it to two doses if stomach upset occurs. This formulation is double distilled and has very little fishy taste, which will make it more palatable for children and will make creating a matching placebo a simpler process.
  Other Names: Nutra Sea HP
  Arms: Omega-3 Fatty Acids
Dietary Supplement: Placebo — Children will be administered 3.75ml of the liquid formulation of Placebo. The starting dose will be 1.875ml and the dose will be doubled on week 2. The parents may choose to give this as a single dose or split it to two doses if stomach upset occurs. This formulation is double distilled and has very little fishy taste, which will make it more palatable for children and will make creating a matching placebo a simpler process.
  Other Names: Placebo Comparator
  Arms: Placebo

SUMMARY:
This is a pilot, randomized, placebo-controlled trial of omega-3 fatty acids in autism. Autism, originally described by Kanner in 1943, is among the most severe of neurodevelopmental disorders. It is a Pervasive Developmental Disorder (PDD) affecting social and communicative functions and is also characterized by repetitive behaviors/restricted interests. It is also frequently accompanied by significant aggression, self-injury, irritability and hyperactivity, making care for these individuals an even greater challenge for families or institutional settings. Autism severely impacts the affected individual and family members, causing life-long functional impairment. In this protocol the investigators will use the terms "autism" and "autism spectrum disorder (ASD)" interchangeably to refer to Autistic disorder, Asperger Syndrome and PDD-Not Otherwise Specified (NOS).

DETAILED DESCRIPTION:
Currently risperidone is the only medication approved the by Food and Drug Administration (FDA) for this disorder, and specifically for irritability associated with autism, although not all patients with autism respond to risperidone. No pharmacologic treatments have been approved for use in preschool children, although it is clear that early intervention is associated with improved outcomes. Behavioral and educational therapies play a significant role in the management of autistic symptoms. The history of alternative treatments in autism is notable for the exaggerated benefit of a variety of supplements, such as high dose vitamins (e.g. B6, magnesium), and secretin. The current widespread use of alternative/nutritional supplements to patients with autism without scientifically demonstrated efficacy, underscores the necessity for scientifically sound studies to be conducted. Complementary and alternative medical therapies (CAM) are commonly employed by families of autistic children. Recent surveys have estimated the prevalence of such use to be between 30% and 95% (1,2,3). Omega-3 fatty acids were reported to be used in 28.7% of patients (1). However, only two small case series and a very small randomized study have been reported in this population to date. The investigators propose to conduct a randomized controlled trial of omega-3 fatty acids in preschoolers with ASD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients 2-5 years of age.
2. Meet Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV) criteria. DSM-IV criteria for an autism spectrum disorder, (Autistic disorder, Asperger syndrome or PDD-NOS) will be established by a clinician with expertise with individuals with ASD based on parent interview, Autism Diagnostic Observation Schedule (ADO) and Autism Diagnostic Interview (ADI-R)
3. If already receiving stable non pharmacologic educational, behavioral, dietary and or/ natural health product interventions during the preceding 3 months prior to Screening, will not electively initiate new or modify ongoing interventions for the duration of the study unless the child's condition is worsening or their turn comes up on the treatment waiting list.
4. Have normal physical examination and laboratory test results at Screening. If abnormal, the finding(s) must be deemed clinically insignificant by the Investigator.
5. The parents must be able to speak and understand English sufficiently to allow for the completion of all study assessments.

Exclusion Criteria:

1. Patients born prior to 35 weeks gestational age.
2. Patients with any primary psychiatric diagnosis other than autism at Screening. We are aware the most primary psychiatric disorders are unlikely to be diagnosed in this age group
3. Patients with a medical history of neurological disease, including, but not limited to, epilepsy/seizure disorder (except simple febrile seizures), movement disorder, tuberous sclerosis, fragile X, and any other known genetic syndromes, or known abnormal MRI/structural lesion of the brain.
4. Patients with a medical condition that might interfere with the conduct of the study, confound interpretation of the study results, or endanger their own well-being. Patients with evidence or history of malignancy or any significant hematological, endocrine, cardiovascular (including any rhythm disorder), respiratory, renal, hepatic, or gastrointestinal disease, or coagulation deficits.
5. Patients taking psychoactive medication(s) (e.g.,stimulants, antidepressants, antipsychotics, antiepileptics, anxiolytics, clonidine).
6. Patients that have been off pharmacotherapy for less than 6 weeks.
7. Patients who are participating in another clinical trial
8. Patients on anticoagulants
9. Patients who know that they will initiate or change nonpharmacologic interventions during the course of the study.
10. Patients unable to tolerate venipuncture procedures for blood sampling.
11. Patients taking Omega-3 supplements who have not discontinued treatment for six weeks prior to entering into the study.
12. Patients who have allergies to any of the ingredients in omega-3 (study product) or the placebo.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2010-11; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evdokia Anagnostou, M.D., Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Mankad D, Dupuis A, Smile S, Roberts W, Brian J, Lui T, Genore L, Zaghloul D, Iaboni A, Marcon PM, Anagnostou E. A randomized, placebo controlled trial of omega-3 fatty acids in the treatment of young children with autism. Mol Autism. 2015 Mar 21;6:18. doi: 10.1186/s13229-015-0010-7. eCollection 2015. PMID 25798215

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the hospital clinical database, as well as presentations at local conferences and media. Diagnosis was established using the Diagnostic and Statistical Manual, Fourth Edition for an Autism Spectrum Disorder supported by the Autism Diagnostic Observations Schedule and the Autism Diagnostic Interview - Revised.
Pre-assignment Details: Participants were randomized to the two arms in a 1:1 fashion by the pharmacy, based on a randomization schedule produced by the study biostatistician. They were stratified into one of four strata based on the PDDBI score obtained at screening (four quartiles).
Groups:
- Omega-3 Fatty Acids: Participants started at 0.75 g of EPA + DHA (1.875 ml once a day) of liquid formulation of NutraSea HP.
  If this was well tolerated, the dose was doubled to 1.5 g (3.5 ml) after 2 weeks, as per Health Canada guidelines for maximum dose for this age group.
  The NutraSea HP formulation is a naturally derived fish oil that is extracted, isolated, and processed to contain EPA/DHA in the ratio of 3:1. It has a lemon flavor.
- Placebo: Participants started at 0.75 g (1.875 ml once a day) of liquid formulation of placebo.
  If this was well tolerated, the dose was doubled to 1.5 g (3.5 ml) after 2 weeks, as per Health Canada guidelines for maximum dose for this age group.
  The placebo had the same physical characteristics as the medication (NutraSea HP) but contained refined olive oil and medium chain triglycerides. The placebo has a lemon flavor.
Period: Overall Study
Arm/Group | Omega-3 Fatty Acids | Placebo
Started | 19 | 19
Completed | 15 | 17
Not Completed | 4 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omega-3 Fatty Acids | Placebo | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19 | 19 | 38
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 15 | 13 | 28
Region of Enrollment [Number; unit: participants]
  Canada | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Pervasive Developmental Disorder-Behavioral Inventory (PDDBI) - Autism Composite Score
Description: The PDDBI measures autism symptomology. The autism composite score was used as the primary outcome measure for autism symptom severity.
  PDDBI Autism Composite Scale Range:
  Minimum Range = 10 (lower autism symptom severity) Maximum Range = 100 (higher autism symptom severity)
  The Autism Composite is calculated from the sum of T-scores of the Sensory/Perceptual Approach Behaviours, Ritualisms/Resistance to Change, Social Pragmatic Problems, and Semantic/Pragmatic Problems domains subtracted by the sum of T-scores of the Social Approach Behaviours, and Expressive Language domain then converted into the Autism Composite as a T-score.
  Mean change between baseline and week 24 is reported. A negative change indicates improvement
Time Frame: Baseline and 24 Weeks
Population: 1 participant was dropped from the analysis in the Omega-3 group as there was insufficient data due to early termination.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Omega-3 Fatty Acids | Placebo
Number analyzed (Participants) | 18 | 19
units on a scale | -4.5 [-8.5 to -0.6] | -6.4 [-10.2 to -2.7]
Statistical Analysis 1: Comparison: Omega-3 Fatty Acids vs Placebo; Test type: Superiority or Other; p = 0.5, Mixed Models Analysis

2. Primary Outcome: Change From Baseline in the Behaviour Assessment System for Children (BASC-2) - Externalizing Problems Composite
Description: The BASC-2 externalizing problems composite measures hyperactivity and aggressive behaviours.
  Primary Outcome domain: Externalizing Problems composite
  Externalizing Problems Composite T-Score Range:
  Minimum Range: 10 (lower externalizing problems) Maximum Range: 120 (higher externalizing problems)
  The Externalizing Problems composite is computed from the sum of t-scores from the hyperactivity and aggression subscales then converted into the externalizing problems composite t-score.
  Mean change between baseline and week 24 is reported. A negative change indicates improvement.
Time Frame: Baseline and 24 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Omega-3 Fatty Acids | Placebo
Number analyzed (Participants) | 18 | 19
units on a scale | 3.2 [-0.5 to 6.9] | -3.0 [-6.6 to 0.6]
Statistical Analysis 1: Comparison: Omega-3 Fatty Acids vs Placebo; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis

3. Secondary Outcome: Number of Participants Classified as Responders by the Clinical Global Impression - Improvement (CGI-I)
Description: The CGI-I is a seven-point scale that provides a clinician rating of global improvement and as such is already inherently a measure of change. It requires the clinician to assess the degree to which the participant's illness has improved or worsened relative to a baseline state before the intervention.
  Change is rated as:
  0- Not assessed
  1. Very Much Improved
  2. Much Improved
  3. Minimally Improved
  4. No Change
  5. Minimally Worse
  6. Much Worse
  7. Very Much Worse
  Participants are classified as responders if their CGI-I score was 1 or 2 and non-responders for CGI-I scores of 3 to 7.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: participants classified as responders
Arm/Group | Omega-3 Fatty Acids | Placebo
Number analyzed (Participants) | 18 | 19
participants classified as responders | 12 | 12

4. Secondary Outcome: Change From Baseline in the Vineland Adaptive Behavioral Scales (VABS) - Adaptive Functioning Composite
Description: The VABS is a measure of adaptive behavior in daily settings. Secondary measure domain: The adaptive functioning composite describes an individuals overall functioning
  Adaptive Behaviour Composite Standard Score Range:
  Minimum range: 20 (low adaptive functioning) Maximum range: 160 (high adaptive functioning)
  The adaptive behaviour composite standard score is computed from the sum of standard scores from the communication, daily living skills, socialization and motor skills domains and converted into the adaptive behavior composite standard score.
  Change in the adaptive behaviour composite standard score from baseline to week 24 is reported. Positive change indicates improvement.
Time Frame: Baseline and 24 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Omega-3 Fatty Acids | Placebo
Number analyzed (Participants) | 18 | 19
units on a scale | 2.8 [0.2 to 5.3] | -0.2 [-2.6 to 2.2]
Statistical Analysis 1: Comparison: Omega-3 Fatty Acids vs Placebo; Test type: Superiority or Other; p = 0.09, Mixed Models Analysis

5. Secondary Outcome: Change From Baseline in the Preschool Language Scale (PLS-4) - Total Language
Description: The PLS-4 is a language measure that provides a global assessment of a child's language functioning abilities, receptive and expressive language.
  Secondary outcome measure domain: Total language standard score
  Total Language Standard Score Range:
  Minimum range: 50 (lower language abilities) Maximum range: 150 (higher language abilities)
  The total language standard score is computed from a sum of the auditory comprehension and expressive communication standard scores, then converted into the total language standard score.
  Change of total language standard scores from baseline to week 24 is reported. Positive change indicates improvement
Time Frame: Baseline and 24 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Omega-3 Fatty Acids | Placebo
Number analyzed (Participants) | 18 | 19
units on a scale | 0.7 [-2.7 to 4.1] | -0.6 [-3.7 to 2.6]
Statistical Analysis 1: Comparison: Omega-3 Fatty Acids vs Placebo; Test type: Superiority or Other; p = 0.6, Regression, Linear

ADVERSE EVENTS:
Groups:
- Omega-3 Fatty Acids: Children will be administered 3.75ml of the liquid formulation of NutraSea HP (containing 1.5 gr of EPA+DHA). The starting dose will be 1.875ml (0.75 gr of EPA+DHA) and the dose will be doubled on week 2. The parents may choose to give this as a single dose or split it to two doses if stomach upset occurs. This formulation is double distilled and has very little fishy taste, which will make it more palatable for children and will make creating a matching placebo a simpler process.
  Omega-3 Fatty Acids: Children will be administered 3.75ml of the liquid formulation of NutraSea HP (containing 1.5 gr of EPA+DHA). The starting dose will be 1.875ml (0.75 gr of EPA+DHA) and the dose will be doubled on week 2. The parents may choose to give this as a single dose or split it to two doses if stomach upset occurs. This formulation is double distilled and has very little fishy taste, which will make it more palatable for children and will make creating a matching placebo a simpler process.
Arm/Group | Omega-3 Fatty Acids | Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 19/19 | 19/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega-3 Fatty Acids (N=19) | Placebo (N=19)
Overactivity (Psychiatric disorders) | 3 (3) | 0 (0)
Decreased Energy (General disorders) | 3 (4) | 2 (2)
Social Communicative Intent Loss (Psychiatric disorders) | 1 (1) | 1 (1)
Staring Spell (Psychiatric disorders) | 1 (1) | 0 (0)
Increased Emotional Lability (Psychiatric disorders) | 1 (1) | 2 (3)
Increased Irritability/Anger/Aggression (Psychiatric disorders) | 7 (10) | 2 (4)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Stuttering (Psychiatric disorders) | 1 (1) | 0 (0)
Increased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 6 (7) | 2 (3)
Decreased Dietary Variety (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 3 (6) | 3 (4)
Regurgitation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 8 (9)
Constipation (Gastrointestinal disorders) | 6 (7) | 6 (7)
Eye Swelling (Eye disorders) | 1 (1) | 0 (0)
Nearsightedness (Eye disorders) | 1 (1) | 0 (0)
Eye Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Earache (Ear and labyrinth disorders) | 3 (3) | 0 (0)
Red Eyes (Eye disorders) | 0 (0) | 1 (1)
Nose Bleed (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Tonsillectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (4)
Daytime Wetting (Renal and urinary disorders) | 1 (1) | 0 (0)
Pain on Urination (Renal and urinary disorders) | 0 (0) | 1 (1)
Change in Urine Colour (Renal and urinary disorders) | 0 (0) | 1 (1)
Muscle Aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Right Leg Internal Rotation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Left Knee Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 6 (10) | 9 (9)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4)
Bruising (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Flaky Scalp (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 16 (23) | 14 (24)
Fever (Infections and infestations) | 4 (4) | 4 (5)
Ear Infection (Infections and infestations) | 1 (1) | 3 (3)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Skin Infection (Infections and infestations) | 1 (1) | 1 (1)
Hand Mouth Foot Disease (Infections and infestations) | 0 (0) | 1 (2)
Roseola (Infections and infestations) | 0 (0) | 1 (1)
Initial Insomnia (Nervous system disorders) | 5 (6) | 4 (4)
Bronchiolitis (Infections and infestations) | 0 (0) | 3 (3)
Hand Mouth Foot Disease (Infections and infestations) | 0 (0) | 1 (2)
Mid-cycle Insomnia (Nervous system disorders) | 3 (6) | 2 (3)
Early Awakening (Nervous system disorders) | 1 (1) | 0 (0)
Non-restorative Sleep (Nervous system disorders) | 1 (1) | 0 (0)
Nightmares (Nervous system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No